CLINICAL TRIAL: NCT04807439
Title: A U.S. Post-Approval Study of the SYNERGYTM Everolimus-Eluting Platinum Chromium Coronary Stent System Evaluating the SYNERGY XLV (MEGATRON) Stent System
Brief Title: A U.S Post Approval Study Evaluating the SYNERGY XLV (MEGATRON) Stent System
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92226704
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Atherosclerosis; Heart Diseases, Coronary; Coronary Artery Disease; Cardiovascular Diseases
Keywords: Drug-Eluting Stents
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SYNERGY XLV (Megatron) Coronary Stent System: The SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System), manufactured by BSC, is a device/drug combination product comprised of two regulated components: a device (Coronary Stent System) and a drug product (a formulation of everolimus contained in a bioabsorbable polymer coating).
  Interventions: Device: SYNERGY XLV (Megatron) Coronary Stent System

INTERVENTIONS:
Device: SYNERGY XLV (Megatron) Coronary Stent System — The SYNERGY MEGATRON Everolimus-Eluting Platinum Chromium Coronary Stent System is indicated for improving luminal diameter in patients, including those at high risk for bleeding, with diabetes mellitus, with symptomatic heart disease, stable angina, unstable angina, non-ST elevation MI or documented silent ischemia due to atherosclerotic lesions in native coronary arteries >3.50 mm to <5.00 mm in diameter in lesions <28 mm in length.

SUMMARY:
This is a post-market, standard of care, real-world observational study to assess the clinical outcomes of the SYNERGY XLV (MEGATRON) Coronary Stent System for the treatment of subjects with atherosclerotic lesion(s) ≤ 28 mm in length (by visual estimate) in native coronary arteries ≥3.50 mm to ≤5.00 mm in diameter (by visual estimate). This Post Approval study is a cohort associated with the Evolve 4.5/5.0 (SYNERGY LV) Post Approval Study, which is registered under ClinicalTrials.gov ID: NCT03875651.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires treatment with a SYNERGY XLV (Megatron) stent

Exclusion Criteria:

* Planned treatment with a non-SYNERGY stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients include those with atherosclerotic coronary lesions with vessel diameters that can appropriately be treated with a SYNERGY Megatron stent according to the commercially approved SYNERGY IFU and the site's local standard of care.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate | 12 Months
  12-month Target Lesion Failure (TLF) rate, defined as any ischemia driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death.

SECONDARY OUTCOMES:
Clinical endpoints | At Hospital Discharge (typically 1-2 days post index procedure), and at 6 months, 12 months, 2 years
  TLR rate, TLF rate (primary endpoint at 12 months), Target vessel revascularization (TVR) rate, Target vessel failure (TVF) rate, MI (Q-wave and non-Q-wave) rate, Cardiac death rate, Non-cardiac death rate, All death rate, Cardiac death or MI rate, All death or MI rate, All death/MI/TVR rate, Stent thrombosis rates (ARC)
Periprocedural endpoints | At Hospital Discharge (typically 1-2 days post index procedure)
  Technical success rate, Clinical procedural success rate

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Stoler, MD, Principal Investigator — Baylor Heart and Vascular Hospital
Locations (8):
- United States (8):
  - Yale University, New Haven, Connecticut
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - North Kansas City Hospital, Kansas City, Missouri
  - Wake Medical Center, Raleigh, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy: (http://www.bostonscientific.com/en-US/data-sharing-requests.html).